CLINICAL TRIAL: NCT01491217
Title: A Phase I-II Clinical Trial to Determine Recommended Dose and to Assess the Efficacy, Safety and Pharmacokinetic Profile of Oral Paclitaxel(Oraxol®) in Patients With Advanced/Metastatic or Recurrent Gastric Cancer
Brief Title: A Study of Oraxol® in Gastric Cancer Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM-OXL-201
Record Dates: First submitted 2011-12-05; First posted 2011-12-13 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Advanced Metastatic Gastric Cancer; Recurrent Gastric Cancer
Keywords: Oraxol®; oral paclitaxel; paclitaxel; HM30181A; MTD; DLT; RD
MeSH Terms: conditions — Stomach Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Paclitaxel — HM30181AK 15 mg tablet + Paclitaxel 10mg, 30mg capsules

SUMMARY:
The main objectives of this study are to determine the maximum tolerated dose (MTD) and recommend dose (RD) of Oraxol® in Phase I and to determine the objective response rate of Oraxol® in Phase II.

DETAILED DESCRIPTION:
Administration Schedule: 1 cycle of Oraxol® is 28 days and Oraxol® is administrated twice a week, total 6 times per cycle (day 1,2,8,9,15 and 16).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must histologically or cytologically be diagnosed to have an advanced solid cancer. (phaseI)
2. Advanced/metastatic/recurred gastric cancer(PhaseII)
3. ECOG performance status ≤ 2
4. Patients have proper bone marrow, kidney, liver function and patients do not have remarkable dysfunction of heart and lung: WBC≥4000/mm3; Platelet ≥100,000/mm3; Hemoglobin≥9.0g/dL; ANC≥ 1,500 /mm3; Creatinine ≤ 1.5mg/dL; AST/ALT/ALP ≤ 3 X the upper limit of normal; Total bilirubin ≤2.0mg/dL *AST/ALT/ALP ≤ 3 X the upper limit of normal but <5 if liver or bone metastasis is present

Exclusion Criteria:

1. Patients with blood tumor (ex, leukemia), uncontrolled infectious disease, neurologic disorders, metastasis to CNS or ileus (patients requiring non-oral administration of anti-biotics to treat active bacterial infection are nor eligible, but patients can participate in the trial after complete eradication or control of the infection)
2. Patients who have received bone marrow transplant or are to receive bone marrow transplant.
3. Patients who had the medical history of atrial or ventricular arrhythmia or congestive heart failure or received medical treatment for myocardial infarction within 6 months.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2009-05; Primary Completion 2012-03 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Toxicity evaluation (safety evaluation) | DLT will be assessed on 28days of 1 cycle
  Toxicity will be evaluated by medical history, vital signs, physical examination and laboratory tests performed during the screening period (D-28 to D0) and treatment period based on NCI-CTCAE (version 3.0).
Overall response rate(ORR) evaluation | Response will be evaluated every Cycle 2(8weeks)
  It is measured up to confirmation of tumor response(CR, PR)
  Tumor response will be evaluated by RECIST v1.0.

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Jue Bang, MD. Ph.D, Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - National Cancer Center, Goyang
  - Seoul National University Hospital, Seoul

REFERENCES:
- [Derived] Lee KW, Lee KH, Zang DY, Park YI, Shin DB, Kim JW, Im SA, Koh SA, Yu KS, Cho JY, Jung JA, Bang YJ. Phase I/II Study of Weekly Oraxol for the Second-Line Treatment of Patients With Metastatic or Recurrent Gastric Cancer. Oncologist. 2015 Aug;20(8):896-7. doi: 10.1634/theoncologist.2015-0202. Epub 2015 Jun 25. PMID 26112004